CLINICAL TRIAL: NCT02082912
Title: NMDA Receptors in Motor Learning in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andrew Butler, PhD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00035176; UL1TR000454 (NIH)
Record Dates: First submitted 2014-03-05; First posted 2014-03-10 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D-cycloserine (Experimental): Subjects will take D-cycloserine and use the HandMentor Pro for robotic therapy
  Interventions: Drug: D-cycloserine; Device: HandMentor Pro
- Placebo (Active Comparator): Subjects will take a placebo pill and use the HandMentor Pro for robotic therapy
  Interventions: Other: Placebo; Device: HandMentor Pro

INTERVENTIONS:
Drug: D-cycloserine — D-cycloserine 100mg PO twice weekly (Monday and Wednesday) for three weeks
  Other Names: Seromycin
  Arms: D-cycloserine
Other: Placebo — Placebo pill PO twice weekly (Monday and Wednesday) for three weeks
  Arms: Placebo
Device: HandMentor Pro — The HandMentor Pro (Kinetic Muscles Inc.) is a robotic device that has recording electrodes. The device gives feedback during various activities requiring varying levels of wrist control. The main goal of the hand robot is to improve active range of motion about the wrist and fingers and wrist control. The robotic therapy will be done over 3 consecutive weeks for 2 hours each session (days 1, 3, 5, 8, 10, 12, 15, 17 and 19, for 18 hours total).

SUMMARY:
The purpose of this study is to focus on enhancing upper limb recovery in patients post-stroke by using robotic-assisted therapy in combination with a drug to improve learning new motor skills.

DETAILED DESCRIPTION:
Disability after a stroke is common, leaving 65% of patients unable to use their affected hand in daily activities after 6 months. Frequently, these limitations can cause a decreased quality of life. The current standard for intense physical therapy most commonly consists of neurofacilitation techniques and/or task-specific training. Labor-intensive and costly therapy methods are critical barriers to achieving optimal functional outcomes in stroke survivors with motor impairments. Thus, there is a great need to find new ways to enhance the effectiveness of upper limb rehabilitation in patients following stroke.

A promising approach to improving upper extremity motor function utilizing repetitive task practice (RTP) and behavioral shaping along with constraint of the less affected limb is constraint-induced movement therapy (CIMT). Two fundamental limitations of CIMT are the time necessary to deliver and oversee training and the excessive time in which the less affected limb must be constrained. RTP, in the context of CIMT appears to be effective in improving upper extremity motor function of patients with stroke. Alternative approaches such as robotic assisted therapy have been investigated. Recent evidence suggests that improvements in upper-extremity motor function, functional performance in daily tasks and quality of life are seen during a robotic-assisted physical therapy regimen.

Activation of N-methyl-D-aspartate (NMDA) receptors is important for inducing various forms of synaptic plasticity. Application of D-cycloserine (a antibiotic for treating tuberculosis) can enhance certain models of plasticity, such as long-term potentiation. Pharmacologic strategies that enhance NMDA neurotransmission and working memory represent a promising adjuvant therapy in motor rehabilitation of patients after stroke.

The researchers for this study have brought these observations together to generate a working hypothesis that D-cycloserine will enhance certain features of motor learning, information processing speed, episodic and working memory and that this effect can be coupled with physical therapy to facilitate retraining of patients to use impaired limbs to a greater extent and faster than they otherwise might be able to do. The researchers specifically hypothesize that motor (re)learning and cognition can be improved in people with post-stroke hemiparesis by increasing the excitability and synaptic activity of the motor cortex by combining D-cycloserine and robotic-assisted physical therapy.

The purpose of this study is to understand the important factors in rehabilitation therapy that help improve arm function after stroke. This information may help to ultimately reduce disability and improve quality of life in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 95 years
* of either sex
* of diverse ethnic background
* have experienced a single unilateral hemispheric or brainstem stroke 3 or more months prior
* if have experienced more than one stroke, will be accepted only if all strokes are on the same side of the brain, there is no history of a clinical ischemic or hemorrhagic event affecting the other hemisphere, and there is no CT or MRI evidence of more than one a lacune or minor ischemic demyelination affecting the other hemisphere.
* active motions of the wrist and hand: 10 of wrist extension from a relaxed flexed position; 10 of extension of any two digits at any joint, and 10 of thumb extension at either joint. All active motions must be repeated 3 times within one minute.
* passive range of motion: 90 of flexion and abduction and 45 external and internal rotation at the shoulder; 45 elbow supination and pronation; elbow extension limited by no more than 30; wrist extension to at least neutral; and digit extension limited by no more than 30.
* participants will not be required to exhibit any active shoulder or elbow motion
* ability to sit independently for at least 2 minutes
* Mini Mental Status Examination score greater than 24
* Motor Activity Log score less than 3
* Prospective participants who qualify but who have profound postural instability will undergo the intervention while walking with contact guarding or, when feasible, using their leg and more involved arm to propel a wheelchair.
* must have a score below 16 on the Center for Epidemiologic Studies Depression Scale
* must receive a score greater than 25 on the Folstein Mini Mental State Exam.

Exclusion Criteria:

* any history of more than minor head trauma, subarachnoid hemorrhage, dementia or any other neurodegenerative disease, multiple sclerosis, HIV infection, drug or alcohol abuse, serious medical illness, schizophrenia, major refractory depression
* insufficient cardiopulmonary function to participate in low-intensity sustained upper extremity exercise
* severe visual impairment
* pregnancy
* breast feeding
* participation in intensive physical therapy within the prior 12 months
* inability to understand the potential risks and benefits of the study, personally provide informed consent, and understand and cooperate with treatment
* participating in other upper extremity rehabilitation, clinical or experimental, during the course of this trial.
* a score of less than 24 on the Folstein Mini-Mental State Exam
* a score of less than10 on the Boston Naming Test
* a first stroke less than 3 months or more than 48 months prior to the initiation of therapeutic intervention
* less than 18 years old
* clinical judgment of excessive frailty or lack of stamina
* serious uncontrolled medical conditions
* excessive pain in any joint of the more affected extremity that could limit ability to cooperate with the intervention
* passive range of motion less than 45 degrees for: abduction, flexion or external rotation at shoulder, or pronation of forearm
* greater than 30 degrees flexion contracture at any finger joint
* unable to stand independently for 2 min., transfer independently to and from the toilet or perform sit-to-stand
* current participation in other pharmacological or physical intervention studies, or have received injections of anti-spasticity drugs into upper extremity musculature within the past 3 months, or wish to have drugs injected in the foreseeable future
* receiving any anti-spasticity drugs orally at the time of expected participation
* received phenol injections less than 12 months prior to receiving therapy
* contemplating a move from proximity to the treatment site in less than 6 months from the randomization date.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bulter, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Butler AJ, Kallos J, Housley SN, LaPlaca MC, Traynelis SF, Wolf SL. Randomized, Placebo-Controlled, Double-Blind Pilot Study of D-Cycloserine in Chronic Stroke. Rehabil Res Pract. 2015;2015:534239. doi: 10.1155/2015/534239. Epub 2015 Oct 26. PMID 26587287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Center for Rehabilitation Medicine at Emory University in Atlanta, Georgia. Enrollment of participants began in June 2010 and study participation ended in April 2012.
Pre-assignment Details: A total of 124 patients were screened and of these 14 met enrollment criteria and consented to participate in the study.
Groups:
- D-cycloserine: Participants taking D-cycloserine and using the HandMentor Pro for robotic therapy
- Placebo: Participants taking a placebo pill and using the HandMentor Pro for robotic therapy
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only participants that completed the study are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (7.3) | 53.7 (18.4) | 55.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Grip Strength of Affected Hand
Description: Hand-grip strength was assessed using the whole hand and was defined as the average of 3 trials using a calibrated Jamar dynamometer (Jamar Dynamometer, Asimow Engineering Co., Santa Monica, CA), with the elbow flexed to 90º and the forearm in a neutral position. This is the standardized method for measuring hand-grip strength with a Jamar dynamometer recommended by the American Society of Hand Therapists. An increase in values means that grip strength is improving.
Time Frame: Baseline, Day 30
Population: Participants completing the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 7 | 6
Newton
  Baseline | 3.95 (2.96) | 5.72 (3.98)
  Day 30 | 4.90 (3.56) | 8.44 (4.90)

2. Secondary Outcome: Percentage of Stroke Impact Scale (SIS) Categories Meeting Change Criteria
Description: The percentages of Stroke Impact Scale (SIS) physical domain categories meeting criteria for Minimal Clinically Important Difference (MCID) are presented here. The SIS has 59 items in 8 domains of function where respondents rate their degree of difficulty on a 5-point scale, plus a 9th category for stroke recovery (one item, scored from 0 to 100). Scores for each domain are generated so that total scores for each domain range from 0 - 100, where higher scores indicate less difficulty and more recovery. A change of more than 4.5 to 17.8 for the domains was considered a MCID. A higher percentage of SIS categories meeting the MCID criteria indicates increased improvement in that study arm.
Time Frame: Baseline, Day 30
Population: Participants completing the study are included in this analysis.
Measure: Number; unit: percentage of category scores
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 7 | 6
percentage of category scores | 44.4 | 24.1

3. Secondary Outcome: Center for Epidemiologic Studies Depression (CES-D) Scale Score
Description: Depressive symptoms were assessed with the Center for Epidemiologic Studies Depression (CES-D) Scale. The CES-S has 20 items rated on a scale of 0 to 3. Total scores range from 0 to 60 with higher scores indicating more depressive symptoms, and a score of 16 or above indicates depression. Baseline scores are presented in the Outcome Measure Data Table and the impact of the study arm at Day 30 is presented in the statistical analysis section.
Time Frame: Baseline, Day 30
Population: Participants completing the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 7 | 6
units on a scale | 15.1 (6.5) | 9.2 (8.8)
Statistical Analysis 1: Comparison: D-cycloserine vs Placebo; Values represent the time x treatment group interaction; Test type: Superiority; p = 0.651, ANOVA; F statistic = 0.216

4. Secondary Outcome: Display Enhanced Testing for Concussions and Mild Traumatic Brain Injury (mTBI) (DETECT) System Score
Description: Using a computer, helmet with heads-up-display, headphones with audio inputs, and an input unit with two buttons ("Yes" and "No"), the DETECT system combines an immersive environment with neuropsychological tests to assess mTBI. The DETECT software consists of a series of tests evaluating information processing speed, episodic memory, and working memory. Performance is scored based on response type (correct, incorrect, and missing) and response time. Test results are displayed using an internal algorithm that is based on the probability of impairment. Mean baseline z-scores are presented in the Outcome Measure Data Table and the impact of the study arm at Day 30 is presented in the statistical analysis section. A z-score of 0 represents a healthy individual; scores above 0 are the number of standard deviations above the mean, indicating more errors, taking more time, and thus having a higher probability of mild cognitive impairment.
Time Frame: Baseline, Day 30
Population: Participants with complete information for the DETECT measurement are included in this analysis. Two participants had missing values dues to technical issues with the instrument.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 6 | 5
z-score | 10.2 (0.0) | 10.1 (0.1)
Statistical Analysis 1: Comparison: D-cycloserine vs Placebo; Values represent the time x treatment group interaction; Test type: Superiority; p = 0.447, ANOVA; F statistic = 0.633

5. Secondary Outcome: Number of Blocks Moved During the Box and Block Test (BBT) of Affected Arm
Description: Change in functional motor task performance of the arm affected by the stroke was assessed with the Box and Block Test (BBT). The BBT involves dexterous manipulation of objects and voluntary motor control, which improves with upper limb recovery following stroke. The number of blocks moved within 60 seconds are counted. Baseline scores of the mean number of blocks moved are presented in the Outcome Measure Data Table and the impact of the study arm at Day 30 is presented in the statistical analysis section.
Time Frame: Baseline, Day 30
Population: Participants completing the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: blocks per minute
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 7 | 6
blocks per minute | 9.7 (7.9) | 9.6 (6.2)
Statistical Analysis 1: Comparison: D-cycloserine vs Placebo; Values represent the time x treatment group interaction; Test type: Superiority; p = 0.471, ANOVA; F statistic = 0.557

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time each participant consented to take part in the trial through the end of study follow up (30 days). Adverse events for all participants who began the study are presented, regardless of whether or not they finished the study.
Arm/Group | D-cycloserine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes